CLINICAL TRIAL: NCT07304583
Title: Investigation of the Effects of Having Children Listen to the Sound of Water and Watching Videos With Water Sounds Using Virtual Reality on Urination, Fear, and Pain in the Postoperative Period
Brief Title: The Effect of Playing the Sound of Water and Watching Videos With VR on Urination, Fear, and Pain in Post-Op Children
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Esma PEKER, graduate student, Ondokuz Mayıs University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: EPEKER
Record Dates: First submitted 2024-12-31; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Urinary Retention Postoperative
Keywords: Child; Urinary retention; Postoperative
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): A group that will not receive any intervention and will be observed. After surgery, children are told not to hold their urine and are observed. 35 children are evaluated.
- Experimental group-1 (listening to water sound) (Experimental): The group that will listen to the sound of water. After the surgery, children are made to listen to the sound of water and their urination times, fear and pain levels are evaluated. 35 children are evaluated.
  Interventions: Other: Listening to the sound of water
- Experimental group-2 (watching videos with VR glasses) (Experimental): The group will watch a video with the sound of water using virtual reality. After the surgery, children are shown a video with the sound of water using VR glasses to assess their urination, pain, and fear. 35 children are evaluated.
  Interventions: Other: Listening to the sound of water

INTERVENTIONS:
Other: Listening to the sound of water — Urination status will be examined by listening to the sound of water or watching a video with water sound through VR glasses.
  Other Names: Watching videos with mute sound using VR glasses
  Arms: Experimental group-1 (listening to water sound); Experimental group-2 (watching videos with VR glasses)

SUMMARY:
It was aimed to investigate the effects of watching a video with water sound via virtual reality and listening to the sound of water through headphones on urination, fear and pain in children in the post-operative period.

DETAILED DESCRIPTION:
Urinary retention is the inability to urinate despite a full bladder and is a common complication of surgery and anesthesia. Excessive urinary pressure and bladder distension are emergencies that can lead to kidney damage or dysfunction. Various methods are used to prevent urinary retention, including imitating the sound of running water, massaging the bladder, taking a warm bath, and perineal water flow. A literature review found no studies examining the effect of the sound of running water on pain, but found studies on other distraction methods used during painful procedures in children. Therefore, this study aimed to investigate the effects of watching a quiet video and listening to the sound of water in a virtual reality setting on urination, fear, and pain in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being within the specified age range

Exclusion Criteria:

* Not volunteering to participate in the study
* Not being within the specified age range

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Wong Baker Facial Pain Assessment Scale | After the research is completed, approximately 6 months
  This scale will be used to assess the level of pain during urination in children
  before and after surgery. A scoring system of 0-10 will be used. 0 indicates no pain, and 10 indicates the most severe possible pain.

SECONDARY OUTCOMES:
Child Fear Scale | After the research is completed, approximately 6 months
  This scale will measure a child's fear of urination before and after surgery. A score of 0-4 will be given, where 0 represents no fear at all and 4 represents the highest possible level of fear.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Tural Büyük, Principal Investigator — Ondokuz Mayıs Universty
Locations (1):
- Ondokuz Mayıs Universty, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No